CLINICAL TRIAL: NCT01609426
Title: Factors of Steroid Dependency in Idiopathic Nephrotic Syndrome
Acronym: NEPHROVIR-2
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI11021; AOM 11002 (Other: Assistance Publique)
Record Dates: First submitted 2012-04-25; First posted 2012-06-01 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Idiopathic Nephrotic Syndrome
Keywords: Proteinuria; idiopathic; nephrotic syndrome; herpesvirus; epidemiology; immune response; interferon; steroid dependency; nephrotic disease: Idiopathic nephrotic syndrome
MeSH Terms: conditions — Nephrosis, Lipoid; Proteinuria; Nephrotic Syndrome; Herpes Simplex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA Peripheral Blood Mononuclear Cells Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children with idiopathic nephrotic syndrome: children below 16 years of age with a steroid dependent nephrotic syndrome
  Interventions: Genetic: DNA chip dedicated to the pharmacogenetic of steroids

INTERVENTIONS:
Genetic: DNA chip dedicated to the pharmacogenetic of steroids — direct DNA extraction from peripheral blood cells

SUMMARY:
The primary purpose of the study is to identify the factors of steroid dependency in childhood idiopathic nephrotic syndrome. The steroid dependency is defined by a relapse of nephrotic syndrome within the 3 weeks that follow the withdrawal of steroid therapy after the first manifestation. Different clinical and biological factors will be analyzed: age of first manifestation, delay of remission, ethnicity, and preceding viral infection, geolocalization in the Parisian area, genoprevalence of herpes viruses and polymorphisms in the genes involved in the response to steroid therapy.

DETAILED DESCRIPTION:
Patients with a steroid dependent nephrotic syndrome will be compared to those with a non steroid dependent form of nephrotic syndrome at the end of the first manifestation. An additional blood volume will be sampled in patients and controls during a scheduled biological check-up for the initial disease. Genetics factors will be checked using a DNA chips devoted to the response to steroid therapy and viral genome of EBV, CMV, HHV7 will be searched for using PCR reaction in total blood DNA extract.

ELIGIBILITY:
Inclusion Criteria:

* children below 16 years
* first manifestation of nephrotic syndrome
* steroid sensitivity according to the recommendations of the french "pediatric society nephrology"

Exclusion Criteria:

* patients who don't stay in Paris during the study

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any children below 16 years of age with a first manifestation of idiopathic nephrotic syndrome commencing or having commenced in the Paris area
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
define pharmacogenetic factors of steroid dependency | 28.5 months

SECONDARY OUTCOMES:
parameters of the immune response against herpesvirus, specially the cellular production of interferon induced by specific viral peptides | 28.5 months
Dynamic of the epidemiology of idiopathic nephrotic syndrome in the Paris Area | 28.5 months
  Number of participants with idiopathic nephrotic syndrome in Paris Area to determinate if clusters cases exist.
Analysis of cortico-dependence factors | Day 1
  Comparison of polymorphisms of cortico-dependent patients with non- cortico-dependent patients
Analysis of susceptibility factors that generate the appearance of the Idiopathic Nephrotic Syndrome | Day 1
  Comparison of polymorphisms of all patients suffering from the Idiopathic Nephrotic Syndrome, with general population

CONTACTS AND LOCATIONS:
Overall Officials: Georges Deschênes, MD-PhD, Principal Investigator — Assistance Publique
Locations (1):
- APHP Robert-Debré, Department of Pediatric Nephrology, Paris, France